CLINICAL TRIAL: NCT04443556
Title: Effect of Continue Rhomboid Intercostal and Subserratus Plane Block in Thorocotomy
Brief Title: Effect of Continue RISS Block in Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Betul Kozanhan, Ass.Prof., Konya Meram State Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RISS THORACOTOMY
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Pain; Thoracotomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol; Anesthetics, Local; Analgesia, Patient-Controlled

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Rhomboid Intercostal and Subserratus Plane Block (Active Comparator): Standart postoperative analgesia + Continue Rhomboid Intercostal and Subserratus Plane Block
  Interventions: Drug: Tramadol; Other: IV PCA
- Control Group (Other): Standart postoperative analgesia
  Interventions: Other: IV PCA

INTERVENTIONS:
Drug: Tramadol — Before the closure of the thoracotomy, the surgeon will place two catheters through a Tuohy needle into fascial planes for continue the RISS block. First catheter tip will be placed towards the interfascial planes between the rhomboid major and intercostal muscles and the second catheter tip will be placed in subserratus fascial plane. Continue local anesthetics will be injected through the catheters for 48 hours. Also an IV patient-controlled analgesia device containing tramadol will be provided. Tramadol consumptions and postoperative numeric rating scale (NRS) scores for pain will be recorded.
  Other Names: Local anesthetic
  Arms: Group Rhomboid Intercostal and Subserratus Plane Block
Other: IV PCA — An IV patient-controlled analgesia device containing tramadol will be provided. Tramadol consumptions and postoperative numeric rating scale (NRS) scores for pain will be recorded.

SUMMARY:
Thoracotomy is one of the most painful surgery. Acute postoperative pain increases postoperative morbidity and prolongs hospital stay and also may lead to developing a chronic pain syndrome. This study aimed to assess the efficacy of continuous rhomboid intercostal and subserratus plane (RISS) block by inserting a catheter under direct vision for controlling acute thoracotomy pain.

DETAILED DESCRIPTION:
Before the closure of the thoracotomy, the surgeon will place two catheters through a Tuohy needle into fascial planes for continue RISS block. First catheter tip will be place towards the interfascial planes between the rhomboid major and intercostal muscles and the second catheter tip will be place in subserratus fascial plane. Continue local anesthetics will be injected through the catheters for 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age undergoing elective thoracic surgery
* American Society of Anesthesiologists (ASA) physical status I-III grade

Exclusion Criteria:

* Patient refusal
* History of psychiatric and cognitive disorders.
* Patients allergic to the drugs used in the study
* Emergent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
postoperative pain | postoperative 48 hour
  Numeric rating scale (NRS) NRS use numbers to rate pain from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Analgesic consumption | Postoperative 48 hour
  Total opioid consumption after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Konya Education and Training Hospital, Konya, Turkey (Türkiye)